CLINICAL TRIAL: NCT03361098
Title: Combined Effects of SGLT2 Inhibition and GLP-1 Receptor Agonism on Food Intake, Body Weight and Central Satiety and Reward Circuits in Obese T2DM Patients
Brief Title: DECREASE: Dapagliflozin Plus Exenatide on Central REgulation of Appetite in diabeteS typE 2
Acronym: DECREASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, RG IJzerman, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DC2017DECREASE01
Record Dates: First submitted 2017-09-26; First posted 2017-12-04 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: SGLT2 inhibition; dapagliflozin; GLP-1 receptor agonist; exenatide; Central satiety and reward circuits; bodyweight; brain
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants were treated in a double-dummy design. There was no difference in appearance between exenatide and placebo injections, or dapagliflozin and placebo tablets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SGLT2 inhibitor + GLP-1 receptor agonist (Experimental): dapagliflozin 10 mg tablet /day and exenatide twice daily subcutaneous injection (week 1-4; 5 microgram, week 5 -16; 10 microgram)
  Interventions: Drug: Dapagliflozin 10mg; Drug: Exenatide
- GLP-1 receptor agonist (exenatide) and placebo (Active Comparator): GLP-1 receptor agonist exenatide twice daily in combination with placebo dapagliflozin
  Interventions: Drug: Exenatide; Other: placebo dapagliflozin
- SGLT2 inhibitor (dapagliflozin) and placebo (Active Comparator): SGLT2 inhibitor dapagliflozin 10 mg tablet /day in combination with placebo GLP-1 receptor agonist exenatide twice daily
  Interventions: Drug: Dapagliflozin 10mg; Other: placebo exenatide
- double placebo (Placebo Comparator): placebo dapagliflozin and placebo exenatide twice daily
  Interventions: Other: placebo exenatide; Other: placebo dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10mg oral tablet once daily
  Other Names: SGLT2 inhibitor ; Forxiga
  Arms: SGLT2 inhibitor (dapagliflozin) and placebo; SGLT2 inhibitor + GLP-1 receptor agonist
Drug: Exenatide — Exenatide 5 microgram b.i.d. week 1-4 Exenatide 10 microgram b.i.d. week 5-16
  Other Names: GLP-1 receptor agonist ; Byetta
  Arms: GLP-1 receptor agonist (exenatide) and placebo; SGLT2 inhibitor + GLP-1 receptor agonist
Other: placebo exenatide — placebo b.i.d. exenatide
  Arms: SGLT2 inhibitor (dapagliflozin) and placebo; double placebo
Other: placebo dapagliflozin — placebo tablets dapagliflozin
  Arms: GLP-1 receptor agonist (exenatide) and placebo; double placebo

SUMMARY:
This is a 16 week, phase 4, randomized and placebo controlled trial, investigating the separate and combined effects of Sodium Glucose coTransporter 2 (SGLT2) inhibition with dapagliflozin and Glucagon Like peptide-1 (GLP-1) receptor agonism with exenatide on food intake, body weight and the neural activity in the central satiety and reward circuits in response to food-related stimuli by blood oxygen level-dependent (BOLD) fMRI in obese type 2 diabetes patients. The investigators hypothesize that treatment with SGLT2 inhibitors is associated with alterations in central reward and satiety circuits in response to food related stimuli, leading to increased appetite and food intake. In addition, the investigators hypothesize that adding a GLP-1 receptor agonist to the treatment with an SGLT2 inhibitor may increase weight loss and prevent the increased food intake during treatment with SGLT2 inhibitors due to effects on neuronal activity of central satiety and reward circuits in response to food-related stimuli in obese patients with T2DM.

DETAILED DESCRIPTION:
The aim of this study is to investigate 1) the seperate and 2) combined actions of SGLT2 inhibition and GLP-1 receptor agonism on food intake, body weight and the activity within the central satiety and reward circuits in response to food-related stimuli and 3) wheter the combination with a GLP-1 receptor agonist can prevent the increased intake observed with SGLT2- inhibition treatment.

Methods: In four groups of obese patients with T2DM (n=16 per group), food intake and neuronal activity in relevant CNS circuits in response to food-related stimuli (using fMRI) will be investigated during 16 week treatment in a double blind placebo-controlled randomized trial with:1) SGLT2 inhibitor dapagliflozin 10 mg/day in combination with placebo GLP-1 receptor agonist exenatide twice daily, 2) GLP-1 receptor agonist exenatide twice daily in combination with placebo dapagliflozin, 3) combination of dapagliflozin 10 mg/day and exenatide twice daily, or 4) placebo dapagliflozin and placebo exenatide twice daily. To correlate changes in brain activity with subsequent feeding behavior, the investigators will measure food intake, self-reported hunger, satiety and mood, during a choice-buffet after the scanning.

Expected results: This project will gain insight into the CNS mechanisms underlying the the effects of seperate and combined treatment with SGLT2 inhibition and GLP-1 receptor agonism. Furthermore, this project will provide insight if combined treatment with a GLP-1 receptor agonist will prevent the increased intake, observed by treatment with an SGLT2 inhibitor, and if so, in the underlying (CNS) mechanisms. These findings may increase the understanding of the development of obesity and weight loss problems in obese and T2DM patients and may support the development of a balanced SGLT2 inhibitor/GLP-1 receptor agonist combination as a treatment strategy for obesity and T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* BMI 27-40 kg/m2
* Stable bodyweight (<5% reported change during the previous 3 months).
* Diagnosed with T2DM > 3 months prior to screening
* Treatment with metformin and/or sulphonylurea at a stable dose for at least 3 months.
* HbA1c 7.0-10% for patients treated with metformin
* HbA1c 7.5-10% for patients treated with metformin and/ or sulphonylurea
* For women: post menopausal (excluding possible menstruation cycle effects)

Exclusion Criteria:

* GLP-1 based therapies, DDP-4 inhibitors, SGLT-2 inhibitors, thiazolidinediones or insulin within 3 months before screening
* Weight-lowering agents within 3 months before screening.
* Congestive heart failure (NYHA II-IV)
* Chronic renal failure (glomerular filtration rate < 45 mL/min/1.73m2 per Modification of Diet in Renal Disease (MDRD))
* Liver disease
* History of gastrointestinal disorders (including gastroparese, pancreatitis and cholelithiasis)
* Patients with MEN2 syndrome or history or family history of medullary thyroid carcinoma
* Neurological illness
* Malignancy (except for basal cell carcinoma)
* History of major heart disease
* History of major renal disease
* Pregnancy or breast feeding
* Implantable devices
* Substance abuse
* Addiction
* Alcohol abuse (defined as: for men > 21 units/week, for women >14 units/week)
* Smoking/ nicotine abuse (defined as: daily smoking / a daily use of nicotine)
* Contra-indication for MRI, such as claustrophobia or pacemaker
* psychiatric illnesses; mood disorders, eating disorders, anxiety disorders, schizophrenia and other psychotic disorders, dissociative disorders, somatoform disorders, delirium, dementia and other cognitive disorders
* Chronic use of centrally acting agents or glucocorticoids within 2 weeks immediately prior to screening
* Use of cytostatic or immune modulatory agents
* History of allergy for exenatide or other GLP-1 RA
* Participation in other studies
* Individuals who have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Individuals who have previously completed or withdrawn from this study or any other study investigating GLP-1 receptor agonist or dipeptidyl peptidase (DPP)-4 within 6 months
* Visual disability, not correctable with glasses or contact lens
* Individuals who, in the opinion of the investigator, are unsuitable in any other way to participate in this study
* Poor commandment of the Dutch language or any (mental) disorder that precludes full understanding the purpose, instruction and hence participation in the study
* Further exclusion criteria will be in compliance with the EMeA SPC of exenatide and dapagliflozin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Differences in neuronal activity in the central reward and satiety circuits in response to food-related stimuli by BOLD fMRI signal | at baseline, after 10 days and after 16 weeks
  Differences in neuronal activity in the central reward and satiety circuits in response to food related stimuli by BOLD fMRI signal compared to baseline and 16 weeks of treatment between the exenatide + dapagliflozine, exenatide +placebo, dapagliflozin+placebo and double placebo arms.

SECONDARY OUTCOMES:
Differences in neuronal activity in the central reward and satiety circuits in response to food-related stimuli by BOLD fMRI signal | at baseline, after 10 days and after 16 weeks
  Differences in neuronal activity in the central reward and satiety circuits in response to food related stimuli by BOLD fMRI signal compared to baseline and 1.5 weeks of treatment and 1.5 and 16 weeks of treatment between the exenatide + dapagliflozine, exenatide +placebo, dapagliflozin+placebo and double placebo arms.
Feeding behaviour; ad libitum lunch buffet | at baseline, after 10 days and after 16 weeks
  Feeding behaviour, measured as quantitative (kcal) changes in food choice, during an ad libitum lunch buffet will be compared between the groups (at baseline and 1,5 week, baseline and 16 weeks and 1.5 and 16 weeks of treatment)
Feeding behaviour; ad libitum lunch buffet | at baseline, after 10 days and after 16 weeks
  Feeding behaviour, measured as qualitative (energy density as well as nutrient composition;carbohydrate/fat/protein) changes in food choice, during an ad libitum lunch buffet will be compared between the groups (at baseline and 1,5 week, baseline and 16 weeks and 1.5 and 16 weeks of treatment)
Self-reported hunger | at baseline, after 10 days and after 16 weeks
  Self-reported hunger, satiety and fullness and prospective food consumption will be rated on 100 mm visual analogue scales before and after the meal
Difference in resting energy expenditure measured by indirect calorimetry measurements | at baseline, after 10 days and after 16 weeks
  Difference in resting energy expenditure measured by indirect calorimetry measurements between the groups (baseline and 16 weeks, baseline and 1.5 weeks and 1.5 and 16 weeks of treatment)
Change in bodyweight (kg) and body mass index (kg/m2) | at baseline, after 10 days and after 16 weeks
  Change in bodyweight (kg) and body mass index (kg/m2) between the groups ( at baseline and 1,5 week, baseline and 16 weeks, 1.5 week and 16 weeks)
Difference in bodycomposition measured by bio electrical impedance analysis and waist and hip circumference measurements (cm) | at baseline, after 10 days and after 16 weeks
  Difference in bodycomposition measured by bio electrical impedance analysis and waist and hip circumference measurements (cm) between the groups (0-1.5, 0-16, 1.5-16)
Difference in resting brain activity by fMRI resting state measurements | at baseline, after 10 days and after 16 weeks
  Difference in resting brain activity by fMRI resting state measurements between groups (0-1.5, 0-16, 1.5-16)
Effect on cardiovascular autonomic balance by cardiovascular reflex test with finger plethysmography (Nexfin) | at baseline, after 10 days and after 16 weeks
  Effect on cardiovascular autonomic balance by cardiovascular reflex test with finger plethysmography (Nexfin) measuring bloodpressure, hartfrequency, ECG between the groups (0-16, 0-1.5, 1.5-16)
Arterial stiffness: Pulse Wave analysis | at baseline, after 10 days and after 16 weeks
  Arterial stiffness: Pulse Wave analysis will be assessed using the Sphygmocor system, a non-invasive system using applanation tonometry between the groups (0-16, 0-1.5, 1.5-16)
Renal measurements collecting 24 hour urine | at baseline, after 10 days and after 16 weeks
  Renal measurements collecting 24 hour urine; glucose excretion (0-1.5, 0-16, 1.5-16), creatinine clearance (0-1.5, 0-16, 1.5-16), tubular function; sodium excretion and urinary pH (0-1.5, 0-16, 1.5-16), renal damage markers albumin/creatinine ratio (0-1.5, 0-16, 1.5-16)
Laboratory parameters | at baseline, after 10 days and after 16 weeks
  Change in the plasma/serum biomarkers of metabolism, liver function, estimated renal function (eGFR), electrolytes, and haematocrit

OTHER OUTCOMES:
Safety outcomes; Adverse events | +/- 21 weeks
  Occurence of adverse events (as reported by the patient) starting at the informed consent untill 30 days after administration of the last dose of study medication
Safety outcome; vital signs | 16 weeks
  Vital signs: pulse rate, bloodpressure, body temperature
Exploratory objective: Cerebral perfusion assessed by Arterial Spin Labeling | 16 weeks
  Cerebral perfusion assessed by Arterial Spin Labeling between groups (0-1.5,0-16, 1.5-16)
Exploratory objective: measurement of hormones | 16 weeks
  blood will be collected to have the opportunity to perform measurements of hormones such as leptin, cortisol, ghrelin.
Exploratory: Microbiome | Baseline and after 16 weeks
  Fecal samples will be collected to determine the (change) microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Richard G IJzerman, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VU Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results, after de-identification
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 3 months and ending 2 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] van Bloemendaal L, Ijzerman RG, Ten Kulve JS, Barkhof F, Diamant M, Veltman DJ, van Duinkerken E. Alterations in white matter volume and integrity in obesity and type 2 diabetes. Metab Brain Dis. 2016 Jun;31(3):621-9. doi: 10.1007/s11011-016-9792-3. Epub 2016 Jan 27. PMID 26815786
- [Background] Ten Kulve JS, Veltman DJ, van Bloemendaal L, Groot PF, Ruhe HG, Barkhof F, Diamant M, Ijzerman RG. Endogenous GLP1 and GLP1 analogue alter CNS responses to palatable food consumption. J Endocrinol. 2016 Apr;229(1):1-12. doi: 10.1530/JOE-15-0461. Epub 2016 Jan 14. PMID 26769912
- [Background] Ten Kulve JS, van Bloemendaal L, Balesar R, IJzerman RG, Swaab DF, Diamant M, la Fleur SE, Alkemade A. Decreased Hypothalamic Glucagon-Like Peptide-1 Receptor Expression in Type 2 Diabetes Patients. J Clin Endocrinol Metab. 2016 May;101(5):2122-9. doi: 10.1210/jc.2015-3291. Epub 2015 Dec 16. PMID 26672638
- [Background] ten Kulve JS, Veltman DJ, van Bloemendaal L, Barkhof F, Deacon CF, Holst JJ, Konrad RJ, Sloan JH, Drent ML, Diamant M, IJzerman RG. Endogenous GLP-1 mediates postprandial reductions in activation in central reward and satiety areas in patients with type 2 diabetes. Diabetologia. 2015 Dec;58(12):2688-98. doi: 10.1007/s00125-015-3754-x. Epub 2015 Sep 18. PMID 26385462
- [Background] van Bloemendaal L, Veltman DJ, ten Kulve JS, Drent ML, Barkhof F, Diamant M, IJzerman RG. Emotional eating is associated with increased brain responses to food-cues and reduced sensitivity to GLP-1 receptor activation. Obesity (Silver Spring). 2015 Oct;23(10):2075-82. doi: 10.1002/oby.21200. Epub 2015 Aug 31. PMID 26331843
- [Background] van Bloemendaal L, Veltman DJ, Ten Kulve JS, Groot PF, Ruhe HG, Barkhof F, Sloan JH, Diamant M, Ijzerman RG. Brain reward-system activation in response to anticipation and consumption of palatable food is altered by glucagon-like peptide-1 receptor activation in humans. Diabetes Obes Metab. 2015 Sep;17(9):878-86. doi: 10.1111/dom.12506. Epub 2015 Jul 22. PMID 26094857
- [Background] van Bloemendaal L, IJzerman RG, Ten Kulve JS, Barkhof F, Konrad RJ, Drent ML, Veltman DJ, Diamant M. GLP-1 receptor activation modulates appetite- and reward-related brain areas in humans. Diabetes. 2014 Dec;63(12):4186-96. doi: 10.2337/db14-0849. Epub 2014 Jul 28. PMID 25071023
- [Background] van Bloemendaal L, Ten Kulve JS, la Fleur SE, Ijzerman RG, Diamant M. Effects of glucagon-like peptide 1 on appetite and body weight: focus on the CNS. J Endocrinol. 2014 Mar 7;221(1):T1-16. doi: 10.1530/JOE-13-0414. Print 2014 Apr. PMID 24323912
- [Background] Devenny JJ, Godonis HE, Harvey SJ, Rooney S, Cullen MJ, Pelleymounter MA. Weight loss induced by chronic dapagliflozin treatment is attenuated by compensatory hyperphagia in diet-induced obese (DIO) rats. Obesity (Silver Spring). 2012 Aug;20(8):1645-52. doi: 10.1038/oby.2012.59. Epub 2012 Mar 8. PMID 22402735
- [Background] Ferrannini G, Hach T, Crowe S, Sanghvi A, Hall KD, Ferrannini E. Energy Balance After Sodium-Glucose Cotransporter 2 Inhibition. Diabetes Care. 2015 Sep;38(9):1730-5. doi: 10.2337/dc15-0355. Epub 2015 Jul 15. PMID 26180105
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Lundkvist P, Pereira MJ, Katsogiannos P, Sjostrom CD, Johnsson E, Eriksson JW. Dapagliflozin once daily plus exenatide once weekly in obese adults without diabetes: Sustained reductions in body weight, glycaemia and blood pressure over 1 year. Diabetes Obes Metab. 2017 Sep;19(9):1276-1288. doi: 10.1111/dom.12954. Epub 2017 May 31. PMID 28345814
- [Background] Frias JP, Guja C, Hardy E, Ahmed A, Dong F, Ohman P, Jabbour SA. Exenatide once weekly plus dapagliflozin once daily versus exenatide or dapagliflozin alone in patients with type 2 diabetes inadequately controlled with metformin monotherapy (DURATION-8): a 28 week, multicentre, double-blind, phase 3, randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Dec;4(12):1004-1016. doi: 10.1016/S2213-8587(16)30267-4. Epub 2016 Sep 16. PMID 27651331
- [Background] Frank S, Laharnar N, Kullmann S, Veit R, Canova C, Hegner YL, Fritsche A, Preissl H. Processing of food pictures: influence of hunger, gender and calorie content. Brain Res. 2010 Sep 2;1350:159-66. doi: 10.1016/j.brainres.2010.04.030. Epub 2010 Apr 25. PMID 20423700
- [Background] Rothemund Y, Preuschhof C, Bohner G, Bauknecht HC, Klingebiel R, Flor H, Klapp BF. Differential activation of the dorsal striatum by high-calorie visual food stimuli in obese individuals. Neuroimage. 2007 Aug 15;37(2):410-21. doi: 10.1016/j.neuroimage.2007.05.008. Epub 2007 May 18. PMID 17566768
- [Background] Rajeev SP, Cuthbertson DJ, Wilding JP. Energy balance and metabolic changes with sodium-glucose co-transporter 2 inhibition. Diabetes Obes Metab. 2016 Feb;18(2):125-34. doi: 10.1111/dom.12578. Epub 2015 Dec 10. PMID 26403227
- [Background] Muskiet MH, Tonneijck L, Smits MM, Kramer MH, Heerspink HJ, van Raalte DH. Pleiotropic effects of type 2 diabetes management strategies on renal risk factors. Lancet Diabetes Endocrinol. 2015 May;3(5):367-81. doi: 10.1016/S2213-8587(15)00030-3. PMID 25943756
- [Background] Muskiet MHA, Tonneijck L, Smits MM, van Baar MJB, Kramer MHH, Hoorn EJ, Joles JA, van Raalte DH. GLP-1 and the kidney: from physiology to pharmacology and outcomes in diabetes. Nat Rev Nephrol. 2017 Oct;13(10):605-628. doi: 10.1038/nrneph.2017.123. Epub 2017 Sep 4. PMID 28869249
- [Background] Murdaugh DL, Cox JE, Cook EW 3rd, Weller RE. fMRI reactivity to high-calorie food pictures predicts short- and long-term outcome in a weight-loss program. Neuroimage. 2012 Feb 1;59(3):2709-21. doi: 10.1016/j.neuroimage.2011.10.071. PMID 22332246
- [Derived] van Ruiten CC, Smits MM, Kok MD, Serne EH, van Raalte DH, Kramer MHH, Nieuwdorp M, IJzerman RG. Mechanisms underlying the blood pressure lowering effects of dapagliflozin, exenatide, and their combination in people with type 2 diabetes: a secondary analysis of a randomized trial. Cardiovasc Diabetol. 2022 Apr 28;21(1):63. doi: 10.1186/s12933-022-01492-x. PMID 35484607
- [Derived] van Ruiten CC, Veltman DJ, Schrantee A, van Bloemendaal L, Barkhof F, Kramer MHH, Nieuwdorp M, IJzerman RG. Effects of Dapagliflozin and Combination Therapy With Exenatide on Food-Cue Induced Brain Activation in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2022 May 17;107(6):e2590-e2599. doi: 10.1210/clinem/dgac043. PMID 35134184